CLINICAL TRIAL: NCT00134602
Title: An Intervention to Promote Adherence to Antiretroviral Medications Among HIV-infected Children 5-12 Years of Age
Brief Title: Pediatric Impact: Promoting Adherence to Medications Among HIV-infected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Jacobi Medical Center (Other); Children's National Research Institute (Other); Howard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-3660; U64/CCU219540; U64/CCU319449
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections
Keywords: HIV infection, antiretroviral therapy, adherence, pediatric
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Needs assessment followed by tailored intervention

SUMMARY:
The purpose of the study is to develop and evaluate an intervention to promote adherence to HIV medications among children 5-12 years of age. It compares changes in antiretroviral (ARV) adherence between the EIG (enhanced intervention group) and an MIG (minimal intervention group) from baseline to 4 months post-intervention.

Secondary outcomes include examining whether improvement in adherence to a medication regimen is associated with improved health outcomes (i.e., viral load, CD4 counts, etc.); identifying and evaluating predictors and/or mediators of adherence; studying the feasibility of electronic recording in measuring adherence in an HIV-infected pediatric population; and evaluating the relationship between the amount of intervention received (i.e., number of hours/number of sessions) and changes in adherence.

DETAILED DESCRIPTION:
The objective of this research is to develop and evaluate an intervention to promote adherence to HIV-medications among children aged 5-12 years. The research will be conducted at Jacobi Medical Center in the Bronx, NY; Children's National Medical Center in Washington, DC; and at Howard University Hospital in Washington, DC. The research will employ a randomized case control study design. Participants (dyads composed of an HIV-infected child and his/her primary caregiver) will be recruited from eligible families within each site's HIV clinic. After the study is explained and informed consent and assent (where applicable) are obtained, participants will be randomly assigned to either the enhanced intervention group (cases) or the minimal intervention group (controls). Participants assigned to the enhanced intervention group will receive a multi-component intervention, specifically tailored to their family's needs, which includes a maximum of 24 hours of contact conducted over a period of up to 12-weeks, and a 1-3 hour booster session approximately six weeks after the intervention phase is completed.

The enhanced intervention will be coordinated by an onsite Adherence Coordinator (AC) and implemented primarily by the AC or another member of the study staff. Participants assigned to the comparison group will receive a minimal intervention that will consist of an educational video and health education pamphlets about general health. All participants will continue to receive the standard-of-care at their respective sites during the study period. Assessments of all participants will be done at baseline (Assessment A), 1 month (Assessment B), and 4 months (Assessment C) following the intervention. Each assessment will include an interview to collect the following information from families:

* socio-demographic data;
* parental/child report of child's medication taking or adherence (self-reported adherence);
* mental health functioning (of parents and child, using standardized measures);
* HIV (of parents) and medication knowledge (of parents and child);
* medical review of child's hospital chart.

The baseline assessment of adherence to medications will include electronic recording of medication taking via a MEMS® cap done over a four-week period. Ongoing electronic assessment of adherence will occur for the duration of the study. Pharmacy refill data will also be obtained for a portion of the study participants for whom data are available.

ELIGIBILITY:
Inclusion Criteria:

* Families with a child between the ages of 5 and 12 years old who is HIV-infected and who receives care at participating hospitals
* Informed consent for and assent from the child
* Informed consent for the primary caregiver (person responsible for most of the child's medication delivery) must be obtained. The parent/legal guardian must be able to give informed consent and willing to comply with protocol requirements.
* The HIV-infected child must be currently prescribed an antiretroviral therapy regimen.

Exclusion Criteria:

* The child or caregiver cannot respond to self-report questions because of cognitive impairments.
* The child receives home health care in which the home health care aide dispenses all of the child's medication (essentially resulting in directly observed therapy for that child).
* The child and/or the caretaker does not speak English or Spanish.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180
Dates: Start 2003-04; Primary Completion 2007-01 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Improved adherence to antiretroviral treatment regimen

SECONDARY OUTCOMES:
Improved viral load
Improved CD4 count

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wiznia, MD, Principal Investigator — Jacobi Medical Center, Bronx, NY; Tamara Rakusan, MD, Principal Investigator — Children's National Research Institute; Sohail Rana, MD, Principal Investigator — Howard University Hospital, Pediatrics Department
Locations (3):
- United States (3):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Howard University Hospital, Department of Pediatrics, Washington D.C., District of Columbia
  - Jacobi Medical Center, The Bronx, New York